CLINICAL TRIAL: NCT00108927
Title: Improving Diabetes Through Primary Care Translation (IMPACT)
Brief Title: Improving Diabetes in Primary Care (IMPACT)
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Other Study IDs: 1 R18 DK061709 (completed); 1R18DK061709 (NIH)
Record Dates: First submitted 2005-04-20; First posted 2005-04-21 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus; Type 2 Diabetes Mellitus; Hypertension
Keywords: Clinical trial; Diabetes; Quality Improvement
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Behavioral: TRANSLATE

SUMMARY:
The goal of our research program is to successfully translate empirical knowledge regarding diabetes treatment and management into sustainable clinical practice. The study hypothesis is that implementation of a multicomponent intervention will result in meaningful improvement in clinical performance measures at the clinic that include average A1c (Hemoglobin A1c), average systolic blood pressure, and national clinical performance measures at a reasonable cost to the health system.

DETAILED DESCRIPTION:
The focus of the study is on the primary care environment, where the majority of patients with diabetes seek on-going health care. The proposed group-randomized and controlled clinical trial-targeted at 24 primary care clinics-evaluates the effectiveness of the TRANSLATE intervention, a multifaceted diabetes intervention program promoting better comprehensive diabetes management. The intervention begins by evaluating the organizational structures of primary care offices and identifying existing barriers in these small complex systems. A set of nine well-developed intervention components-selected from among some of the most successful strategies in the literature for altering clinical outcomes-are then introduced to correct existing deficiencies at each clinic. The TRANSLATE components function as an interdependent system, providing substantial support to both the provider and patient. Key features include the targeting of high-risk patients, a patient reminder system for routine visits, both passive and patient-specific physician reminders, a disease-specific networked reporting system, and physician education. Implementation is facilitated by a local diabetes intervention team assisted by a site coordinator and a local physician champion. Notably, the model does not centralize care, but rather promotes dissemination of care delivery improvements by promoting infrastructure changes at the primary care clinic where most care is delivered. Quality improvement methods are employed to optimize implementation in each unique clinic setting. Upper level administrative personnel are integrated into the regular review of implementation measures and resource use.

The study hypothesis is that implementation of the TRANSLATE intervention will result in meaningful improvement in physiologic outcome measures and important disease process measures-at a reasonable cost-within primary care settings.

The specific aims of the project are to rigorously evaluate the effectiveness of the TRANSLATE program by comparing intervention and control clinics on the following three clinical and economic outcomes:

1. the change in A1c and systolic blood pressure values among all patients with diagnosed diabetes mellitus in participating primary care clinics over 12 months;
2. the quality of diabetes care delivery as measured by the distribution and prevalence of appropriate A1c, microalbumin, low density lipoprotein measurements, and foot exams over 12 months;
3. the economic impact on the health care delivery system as measured by the short- and long-term cost from the perspective of the health care system.

ELIGIBILITY:
Inclusion Criteria:

(The unit of randomization is the medical clinic)

* Clinics were excluded if they participated in an effective quality improvement program within the last two years.
* Clinics must have 3-22 full time equivalent providers
* Clinics must be located in Minnesota or Western Wisconsin
* Clinics must be willing to implement a diabetes registry
* Must be a single specialty, general internal medicine or family practice clinic

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6000
Dates: Start 2003-12; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Peterson, MD MPH, Principal Investigator — University of Minnesota
Locations (1):
- Dept of Family Medicine and Community Health, University of Minnesota Medical School, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Peterson KA, Radosevich DM, O'Connor PJ, Nyman JA, Prineas RJ, Smith SA, Arneson TJ, Corbett VA, Weinhandl JC, Lange CJ, Hannan PJ. Improving Diabetes Care in Practice: findings from the TRANSLATE trial. Diabetes Care. 2008 Dec;31(12):2238-43. doi: 10.2337/dc08-2034. Epub 2008 Sep 22. PMID 18809622